CLINICAL TRIAL: NCT01019577
Title: Phase II Clinical Study of Ixabepilone (BMS-247550) by Every-3-week Dosing Regimen in Patients With Metastatic Breast Cancer Previously Treated With an Anthracycline and Who Are Taxane Resistant
Brief Title: Clinical Study of Ixabepilone (BMS-247550) by Every-3-week Dosing Regimen in Patients With Metastatic Breast Cancer Previously Treated With an Anthracycline and Who Are Taxane Resistant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-107
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixabepilone (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Lyophilized and solvent, IV, 10-50 mg/m2, Q3W, Maximum 9 cycles
  Other Names: Ixempra; BMS-247550

SUMMARY:
The purpose of this study is to determine the response rates for Ixabepilone (BMS-247550) in subjects with metastatic breast cancer previously treated with an anthracycline and who are taxane resistant.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 years or older
* Patients with metastatic breast cancer whose primary lesion was definitely diagnosed to be breast by histological or cellular examination

Exclusion Criteria:

* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≥ 2

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To assess the tumor response using RECIST Criteria to determine the best overall response and response rate | For a maximum of 9 3-week cycles or until unacceptable toxicity

SECONDARY OUTCOMES:
To evaluate safety of BMS-247550 (AEs, SAEs, Deaths, treatment related AEs) using CTC Criteria | Every cycle
To evaluate the duration of achieved responses | For a maximum of 9 3-week cycles or until unacceptable toxicity
To evaluate time to progression (TTP) | For a maximum of 9 3-week cycles or until unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx